CLINICAL TRIAL: NCT06906055
Title: Below-the-Knee Interventions for Limb Salvage: Use of Multifunctional Angioplasty Balloon Catheters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Summa Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-0119-01
Record Dates: First submitted 2025-02-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease Below the Knee; Peripheral Arterial Disease, Rutherford 4 and 5 with Possibility to Improve Vascularization
Keywords: angioplasty; limb threatening ischemia; amputation; diabetes; chronic kidney disease; ischemic ulcer; rest pain; gangrene; atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus; Renal Insufficiency, Chronic; Gangrene; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Use of conventional single function crossing catheters, diagnostic catheters, angioplasty balloon catheters
  Interventions: Device: Standard of Care (SOC)
- Finesse BTK Multicath (Experimental): Use of a multifunctional revascularization catheter
  Interventions: Device: Multicath

INTERVENTIONS:
Device: Multicath — Use of a multifunctional catheter for revascularization of blocked arteries below the knee
  Arms: Finesse BTK Multicath
Device: Standard of Care (SOC) — Use of single function crossing catheters, diagnostic catheters, angioplasty balloon catheters
  Arms: Standard of care

SUMMARY:
Below-the-Knee Interventions for Limb Salvage: Use of Multifunctional Angioplasty Balloon Catheters ("BTK Multicath Registry")

A non-randomized clinical registry

This study is designed to obtain preliminary data on clinically relevant procedural variables during percutaneous below-knee artery revascularization procedures among consecutive patients treated with either the Finesse BTK Multicath® ("Finesse") or the standard of care using conventional angioplasty balloon catheters.

This registry will enroll participants with a history of chronic limb threatening ischemia and below-knee arterial insufficiency who will be assigned to revascularization with or without use of the Finesse BTK Multicath. The registry is an acute study examining procedural data only. The primary endpoints of interest are the volume of contrast used for the intervention, overall procedure time, radiation dose, number of catheter exchanges during revascularization, and medical device supply costs. For the first phase 12 consecutive patients will be treated with the standard of care. For the second phase 12 consecutive patients will be treated with Finesse.

24 participants total

Up to 5 study sites in the United States

Initial anticipated enrollment: Q4 2024 Last anticipated enrollment: Q2 2025

Patients >=18 years old with documented history of unilateral chronic limb threatening ischemia due to below-knee arterial insufficiency with angiographic runoff in the foot and limited arterial insufficiency above the knee

1. Contrast volume administered during the revascularization portion of a procedure.
2. Number of catheter exchanges during revascularization
3. Fluoroscopy time
4. Radiation dose during revascularization
5. Procedure time post-enrollment
6. Equipment costs
7. Reduced use of supplies
8. Technical success
9. Safety/Major Adverse Peripheral Events

On-treatment sample Intention-to-treat

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide written informed consent prior to any clinical investigation-related procedures.
* Age ≥ 18 years
* Planned lower extremity catheter-based revascularization for Rutherford 4 through 6 chronic limb-threatening ischemia (Table 1)
* Stenotic (>=70% stenosis by visual estimate) or occlusive lesion in an infrapopliteal artery (anterior tibial, peroneal, or posterior tibial) by angiography
* Target lesion up to 25cm in length by angiography

Exclusion Criteria:

* Participation in another clinical investigation that has not yet completed its primary end point.
* Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population.
* Female subjects of childbearing potential unless negative pregnancy test or contraceptive use
* Bilateral critical limb ischemia
* Planned bilateral vascular intervention
* Lack of reconstitution of foot runoff vessels at ankle joint
* Planned below-the-ankle intervention after completion of diagnostic angiography
* Planned suprainguinal intervention ->=5cm with at least 50% stenosis of the above knee femoro-popliteal artery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Contrast volume | during the intervention/procedure/surgery

OTHER OUTCOMES:
Procedure duration | during the intervention
Radiation dose | during the intervention
Fluoroscopy time | during the intervention
Number of catheter exchanges | during the intervention
Equipment costs | during the intervention
Rate of use of microcatheters or diagnostic catheters | during the intervention/procedure/surgery
Rate of technically successful revascularization of a continuous artery in the calf | during the intervention/procedure/surgery
Adverse events | during the intervention

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Endovascular Consultants, Wilmington, Delaware
  - Atlantic Medical Imaging, Vineland, New Jersey

IPD SHARING:
Plan to Share IPD: No